CLINICAL TRIAL: NCT05110326
Title: Comparison of Ergon Technique Versus Proprioceptive Neuromuscular Facilitation Stretching on Hamstring Flexibility in Patients With Knee Osteoarthritis
Brief Title: Ergon Technique Versus PNF Stretching on Hamstring Flexibility in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Narmeen Anjum
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Ergon Technique; Proprioceptive Neuromuscular Facilitation stretching; Active Knee Extension Test; Western Ontario and McMaster Universities Arthritis Index; Visual Analogue Scale
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERGON Technique Group (Experimental): Patients in this group will receive ERGON Technique along with conventional therapy
  Interventions: Other: ERGON Technique
- Proprioceptive Neuromuscular Facilitation(PNF) stretching Group (Experimental): Patients in this group will receive Proprioceptive Neuromuscular Facilitation (PNF) stretching along with conventional therapy
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF) stretching

INTERVENTIONS:
Other: ERGON Technique — * Hot pack for 15 minutes.
  * Patient position: Prone with knee flexion approximately 45◦.
  * Position of therapist: Standing at the affected side of patient.
  * Technique:Massage cream will be applied on the hamstring and overactive or short muscle fibres that are restricted.The instrument will be applied parallel to the muscle fibers, both in a distal to proximal and them proximal to distal direction as needed.Then gentle massage stroking from the origin to the insertion will be performed using the instrument. Instrument Assisted Soft Tissue Mobilization(IASTM) will be applied for 5 minutes.
  * Strengthening exercises for quadriceps and hamstring will then be performed.
  * Isometrics exercises of Quadriceps: By placing a towel roll below the knee and press and hold for 20 seconds, 5 sets.
  * Isometrics exercises Hamstrings: By placing a towel roll below the knee and press and hold for 20 seconds, 5 sets.
  * Wall sits: For 10 seconds, 5 sets.
  Arms: ERGON Technique Group
Other: Proprioceptive Neuromuscular Facilitation (PNF) stretching — * The patient will be laid down prone and moist heat will be given for 15 minutes prior to stretching the hamstrings.
  * Then patient will be lying supine with hip in 90⁰ of flexion. Patient's knee will be extended until a very mild stretching sensation is felt in hamstring muscles.
  * Then patient will be asked to flex the knee against the resistance applied by hand of therapist.
  * The patient will be asked to use a force of around 50% of maximal strength and an isometric form of contraction will be gained in the hamstring muscles. The patient will hold the contraction for 8 seconds and then the therapist command to relax the hamstring muscle.
  * Immediately after the muscle relaxation the therapist further stretches the hamstring muscles up to a point where the subject reported a mild to moderate stretching sensation without any pain and will be held for 30 seconds.
  * The procedure will be repeated 3 times in every session.
  Strengthening Exercises:
  * Same as ERGON Group
  Arms: Proprioceptive Neuromuscular Facilitation(PNF) stretching Group

SUMMARY:
The study will be a randomized control trial and will be conducted in Pakistan Railway Hospital Rawalpindi. A sample of 60 participants will be taken. Patients will be divided into two groups (A&B) of 30 participants in each group by sealed envelope method. Hot pack will be applied to both groups for 15 minutes at the start of intervention. ERGON Technique(IASTM) will be applied to group A along with strengthening exercise. Proprioceptive Neuromuscular Facilitation (PNF) stretching will be given to group B along with strengthening exercise. A 35 minute session will be given to the patients and 3 sessions will be given once a week. Intervention will be given for 6 weeks. The outcome measure will be Visual analog Scale (VAS), Western Ontario and McMaster Universities Arthritis Index (WOMAC), and Active Knee Extension Test (AKE) will be measured at baseline and at the end of 6th week. Data will be analyzed by SPSS 22.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral/bilateral osteoarthritis
* Participants with unilateral/bilateral hamstring tightness
* 200 from Active Knee Extension test
* Grade 1 and 2 in Kellgren and Lawrence criteria for knee osteoarthritis

Exclusion Criteria:

* Participant failing to fall in the category below will be excluded from the study:
* Any lower extremity injury in past 3 months
* Any fracture or surgery done for pelvis, hip or knee.
* Any neurological symptoms.
* Any recent knee reconstructive surgery
* Burns of lower extremities
* Other musculoskeletal disorders associated with knee joint, Iliotibial band, adductor muscle and Sartorius muscle tightness

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 6 Weeks
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain. It is used to find out the intensity of pain.
Western Ontario and McMaster Universities Arthritis Index(WOMAC) | 6 Weeks
  The Western Ontario and McMaster Universities Arthritis Index(WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales.
Active Knee Extension Test | 6 Weeks
  The Active Knee Extension Test is used to assess hamstring muscle length and the range of active knee extension in the position of hip flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- RHS Rehabilitation Centre, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anjum N, Sheikh RK, Omer A, Anwar K, Khan MMH, Aftab A, Awan WA. Comparison of instrument-assisted soft tissue mobilization and proprioceptive neuromuscular stretching on hamstring flexibility in patients with knee osteoarthritis. PeerJ. 2023 Dec 1;11:e16506. doi: 10.7717/peerj.16506. eCollection 2023. PMID 38054019